CLINICAL TRIAL: NCT01346332
Title: Performance of the Iontophoresis System With Headset in Healthy Volunteers
Brief Title: Healthy Volunteer Study
Acronym: IPSHS
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Other Study IDs: CPR005021
Record Dates: First submitted 2011-04-29; First posted 2011-05-03 (Estimated); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia of Tympanic Membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anesthetization
  Interventions: Device: Iontophoresis System with Headset

INTERVENTIONS:
Device: Iontophoresis System with Headset — Iontophoresis of an anesthesia solution to the tympanic membrane using the Acclarent Iontophoresis System with Headset

SUMMARY:
The study will recruit healthy volunteers to undergo the iontophoresis procedure using the Acclarent Iontophoresis System with Headset.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 years old

Exclusion Criteria:

* Pregnant or lactating females
* Subject with a history of sensitivity or reaction to lidocaine, tetracaine, epinephrine, or any hypersensitivity to local anesthetics of the amide type, or any component of the drug solution
* Significant atrophic or perforated tympanic membrane
* Otitis externa
* Damaged or denuded skin in the auditory canal
* Electrically sensitive subjects and subjects with electrically sensitive support systems (pacemakers, defibrillators, etc.)
* Cerumen impaction resulting in a significant amount of cleaning required to visualize the tympanic membrane
* Evidence of Otitis Media at day of procedure, or within the past three (3) months prior to procedure

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2012-02-01 (Actual); Study Completion 2012-02-01 (Actual)

PRIMARY OUTCOMES:
Pain scores on visual analog scale | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Roberson, MD, Principal Investigator — CEI Medical Group
Locations (1):
- CEI Medical Group, East Palo Alto, California, United States